CLINICAL TRIAL: NCT01861847
Title: 7-Keto DHEA for the Treatment of PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Humanetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2905
Record Dates: First submitted 2013-05-10; First posted 2013-05-24 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 7-oxodehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Group (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo
- Drug group (Active Comparator): 7 Keto-DHEA
  Interventions: Drug: 7-Keto Dehydroepiandrosterone

INTERVENTIONS:
Drug: 7-Keto Dehydroepiandrosterone — 7-Keto Dehydroepiandrosterone, 100 mg capsules given orally twice daily for 4 weeks in one of the two intervention phases, dependent on randomization assignment.
  Other Names: 7-Keto DHEA
  Arms: Drug group
Drug: Placebo — Placebo, 100 mg capsules given orally twice daily for 4 weeks in one of the two intervention phases, dependent on randomization assignment.
  Arms: Placebo Group

SUMMARY:
The purpose of this research study is to test the effectiveness of 7-Keto DHEA in reducing symptoms of Post-Traumatic Stress Disorder (PTSD).

DETAILED DESCRIPTION:
The main purpose of the study is to investigate the possible effect of 7-Keto Dehydroepiandrosterone (7-Keto DHEA) on decreasing Post Traumatic Stress Disorder Symptoms (PTSD) in a Veteran population. The study proposes, based on a 2006 report, that the use of the drug will show significant reduction in overall PTSD symptoms, a decrease in physiological stress response and higher patient-reported quality of life compared to placebo. This is a Phase 2, randomized, double-blind, crossover design with a placebo control. The sponsor for this study is Humanetics Corporation

ELIGIBILITY:
Inclusion Criteria:

* Veteran status and enrolled for care in the Veteran Health Administration
* Ages 18-64
* Primary diagnosis of PTSD as assess by the clinician administered PTSD scale and independent clinical mental health evaluation

Exclusion Criteria:

* psychosis
* Dementia
* Active alcohol and/or substance abuse or dependence
* Active suicidal or homicidal ideation
* Medical concerns that would exclude use of 7-Keto DHEA

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Psychological benefits of 7-Keto DHEA (Dehydroepiandrosterone) in Veterans suffering from PTSD participating in the intervention through questionnaires and corresponding measurement of blood work for amounts of DHEA. | Four months
  Outcome measures include analysis in symptoms of depression, anxiety, stress, trauma, and improved memory and cognitive functioning after treatment with 7-Keto DHEA. Measures will include psychological questionnaires as follows:
  PTSD Checklist (PCL-C) Associated Symptoms of PTSD Scale (ASP) Trauma Symptom Inventory (TSI) Dissociative Experience Scale (DES) Beck Depression Inventory - II (BDI-II) Brief Symptom Inventory (BSI) Quality of Life Inventory (QOLI)
Physiological benefits of 7-Keto DHEA (Dehydroepiandrosterone) in Veterans suffering from PTSD participating in the intervention through questionnaires and corresponding measurement of blood work for amounts of DHEA. | Four months
  DHEA (DHEA-S) concentrations (serum, saliva) are often elevated in men and women suffering from PTSD including that related to combat experience. Several studies have shown an association between higher levels of DHEA/DHEA-S and abatement of PTSD symptoms. Outcome measures include analysis of medical assessments via blood work; Complete Blood Count (CBC), Cortisol, and DHEA sulfate level

CONTACTS AND LOCATIONS:
Overall Officials: Alina Gonzalez-Mayo, MD, Principal Investigator — Bay Pines VAHCS
Locations (1):
- Bay Pines VA Healthcare System, Bay Pines, Florida, United States